CLINICAL TRIAL: NCT01461499
Title: Clinical Investigation on the Effects of Reducing Microalbuminuria in Hypertensive Patients With Type 2 Diabetes - SMART2
Brief Title: Shiga Microalbuminuria Reduction Trial-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shiga University (Other)
Responsible Party: Principal Investigator, Hiroshi Maegawa, Professor of Medicine, Shiga University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMART-2
Record Dates: First submitted 2011-10-19; First posted 2011-10-28 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2017-08

CONDITIONS: Type 2 Diabetes Mellitus; Hypertension
Keywords: Hypertension; Albuminuria; Direct renin inhibitor; Angiotensin receptor blocker; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Albuminuria | interventions — aliskiren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Direct renin inhibitor (Active Comparator)
  Interventions: Drug: Aliskiren
- Angiotensin receptor blockers (Active Comparator)
  Interventions: Drug: any angiotensin receptor blockers

INTERVENTIONS:
Drug: Aliskiren — The patient will start taking one a daily 150 mg/day of aliskiren. In case blood pressure doesn't reach the target (SBP/DBP < 130/80 mmHg), higher dose of aliskiren will be given.In case the blood pressure doesn't achieve the target, another anti-hypertensive drug other than RAS inhibitors (ARB or ACE-inhibitor) or potassium-retaining diuretics will be added from the minimum effective dose.
  Arms: Direct renin inhibitor
Drug: any angiotensin receptor blockers — The patient will start taking one a standard dose of an ARB in Japan. In case blood pressure doesn't reach the target (SBP/DBP < 130/80 mmHg), higher dose of the ARB will be given. In case the blood pressure doesn't achieve the target, another anti-hypertensive drug other than RAS inhibitors (DRI, another ARB or ACE-inhibitor) or potassium-retaining diuretics will be added from the minimum effective dose.
  Arms: Angiotensin receptor blockers

SUMMARY:
The purpose of this study is to compare the effects of a direct renin inhibitor (DRI), aliskiren, on the urinary albumin excretion in hypertensive patients with type 2 diabetes under strict blood pressure control with angiotensin receptor blocker (ARB).

ELIGIBILITY:
Inclusion Criteria:

* Segment: outpatients
* Hypertension: taking an anti-hypertensive treatment or indicating mean sitting SBP/DBP more than130/80 mmHg
* Type 2 diabetes: diagnosed by ADA criteria or under an anti-diabetic drug treatment
* Microalbuminuria: 10 < and < 300 mg/gCr
* Informed consent: patients who understand well about this study based on own voluntary will and can give a written consent

Exclusion Criteria:

* Sever hypertension (over 180/110 mmHg), malignant hypertension and secondary hypertension
* Type 1 diabetes
* Patients whose investigator regards as difficult to comply with study protocol in reference to the package insert of aliskiren
* Patients who have history of operation in gastrointestinal tract surgery, and anamnestic or concurrent gastrointestinal disorders, which may interfere with drug absorption
* Serum potassium > 5.6 mEq/L (hyperkalemia)
* Urinary microalbumin < 10 or > 300 mg/gCr
* Patients who participated in another clinical study within three months

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2011-10; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Maegawa, M.D., Study Chair — Shiga University of Medical Science
Locations (1):
- Shiga University of Medical Science, Ōtsu, Shiga, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Direct Renin Inhibitor: Aliskiren:
  A total of 119 patients were randomly assigned to receive direct renin inhibitor. Eight patients dropped out during the observation period and a total of 111 patients were studied in this group.
- Angiotensin Receptor Blockers: A total of 118 patients were randomly assigned to receive angiotensin receptor blockers. Four patients dropped out during the observation period and a total of 114 patients were studied in this group.
Period: Overall Study
Arm/Group | Direct Renin Inhibitor | Angiotensin Receptor Blockers
Started | 119 | 118
Completed | 111 | 114
Not Completed | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Direct Renin Inhibitor | Angiotensin Receptor Blockers | Total
Number analyzed (Participants) | 111 | 114 | 225
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 57 | 112
  >=65 years | 56 | 57 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (9.3) | 63.0 (8.4) | 63.0 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 33 | 67
  Male | 77 | 81 | 158
Region of Enrollment [Number; unit: participants]
  Japan | 111 | 114 | 225

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Albuminuria
Description: Change in the urinary albumin to creatinine ratio (UACR) from the baseline
Time Frame: baseline and 24 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of UACR change
Groups:
- Direct Renin Inhibitor: Aliskiren: The patient will start taking one a daily 150 mg/day of aliskiren. In case blood pressure doesn't reach the target (SBP/DBP < 130/80 mmHg), higher dose of aliskiren will be given.In case the blood pressure doesn't achieve the target, another anti-hypertensive drug other than RAS inhibitors (ARB or ACE-inhibitor) or potassium-retaining diuretics will be added from the minimum effective dose.
  A total of 378 patients were enrolled for screening, and 141 were not meeting inclusion criteria. Thus, 237 were randomly assigned to receive either direct renin inhibitor (119) or angiotensin receptor blockers (118). Eight patients dropped out during the observation period and a total of 111 patients were studied in this group.
- Angiotensin Receptor Blockers: any angiotensin receptor blockers: The patient will start taking one a standard dose of an ARB in Japan. In case blood pressure doesn't reach the target (SBP/DBP < 130/80 mmHg), higher dose of the ARB will be given. In case the blood pressure doesn't achieve the target, another anti-hypertensive drug other than RAS inhibitors (DRI, another ARB or ACE-inhibitor) or potassium-retaining diuretics will be added from the minimum effective dose.
  A total of 378 patients were enrolled for screening, and 141 were not meeting inclusion criteria. Thus, 237 were randomly assigned to receive either direct renin inhibitor (119) or angiotensin receptor blockers (118). Four patients dropped out during the observation period and a total of 114 patients were studied in this group.
Arm/Group | Direct Renin Inhibitor | Angiotensin Receptor Blockers
Number analyzed (Participants) | 111 | 114
percentage of UACR change | -5.5 [-13.5 to 2.5] | -6.7 [-20.3 to 0.6]

2. Secondary Outcome: Change in the Urinary Angiotensinogen Level
Description: Change in the urinaryurinary angiotensinogen level from the baseline
Time Frame: baseline and 24 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of change UATGCR
Groups:
- Direct Renin Inhibitor: Aliskiren:
  A total of 378 patients were enrolled for screening, and 141 were not meeting inclusion criteria. Thus, 237 were randomly assigned to receive either direct renin inhibitor (119) or angiotensin receptor blockers (118). Eight patients dropped out during the observation period and a total of 111 patients were studied in this group.
- Angiotensin Receptor Blockers: Angiotensin receptor blockers: A total of 378 patients were enrolled for screening, and 141 were not meeting inclusion criteria. Thus, 237 were randomly assigned to receive either direct renin inhibitor (119) or angiotensin receptor blockers (118). Four patients dropped out during the observation period and a total of 114 patients were studied in this group.
Arm/Group | Direct Renin Inhibitor | Angiotensin Receptor Blockers
Number analyzed (Participants) | 111 | 114
percentage of change UATGCR | -1.7 [-10.4 to 7.9] | -5.4 [-22.1 to 1.6]

3. Secondary Outcome: Change in the Plasma Renin Activity
Time Frame: baseline and 24 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Change in the Serum Insulin Level
Time Frame: baseline and 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Direct Renin Inhibitor: Aliskiren: The patient will start taking one a daily 150 mg/day of aliskiren. In case blood pressure doesn't reach the target (SBP/DBP < 130/80 mmHg), higher dose of aliskiren will be given.In case the blood pressure doesn't achieve the target, another anti-hypertensive drug other than RAS inhibitors (ARB or ACE-inhibitor) or potassium-retaining diuretics will be added from the minimum effective dose.
  378 patients were enrolled for screening, and 237 were randomly assigned to receive either direct renin inhibitor (119) or angiotensin receptor blockers (118). Eight patients dropped out during the observation period and a total of 111 patients were studied in this group.
- Angiotensin Receptor Blockers: any angiotensin receptor blockers: The patient will start taking one a standard dose of an ARB in Japan. In case blood pressure doesn't reach the target (SBP/DBP < 130/80 mmHg), higher dose of the ARB will be given. In case the blood pressure doesn't achieve the target, another anti-hypertensive drug other than RAS inhibitors (DRI, another ARB or ACE-inhibitor) or potassium-retaining diuretics will be added from the minimum effective dose.
  378 patients were enrolled for screening, and 237 were randomly assigned to receive either direct renin inhibitor (119) or angiotensin receptor blockers (118). Four patients dropped out during the observation period and a total of 114 patients were studied in this group.
Arm/Group | Direct Renin Inhibitor | Angiotensin Receptor Blockers
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/118
Serious Adverse Events (participants affected / at risk) | 0/119 | 0/118
Other Adverse Events (participants affected / at risk) | 2/119 | 2/118
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Direct Renin Inhibitor (N=119) | Angiotensin Receptor Blockers (N=118)
pneumonia (Infections and infestations) | 2 (5) | 2 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No